CLINICAL TRIAL: NCT05411900
Title: BotulInum Toxin Type A for Peripheral Neuropathic Pain in subjEcts With Carpal Tunnel Syndrome: a Multicenter, Randomized, Doubleblind, Placebo-controlled Study
Brief Title: BotulInum Toxin Type A for Peripheral Neuropathic Pain in subjEcts With Carpal Tunnel Syndrome
Acronym: INjECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Francesco Bono (Other)
Responsible Party: Sponsor-Investigator, Francesco Bono, Principal Investigator, Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
Organization: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT number 2021-006048-29
Record Dates: First submitted 2022-05-27; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Carpal Tunnel Syndrome; Neurogenic Inflammation; Pain; Drug Use; Neuropathic Pain
Keywords: Quality of life; Neuropathic Pain; Botulinum toxin type A; Paroxysmal pain; Carpal tunnel syndrome; Safety
MeSH Terms: conditions — Carpal Tunnel Syndrome; Neurogenic Inflammation; Pain; Neuralgia | interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Interventional prospective, multicenter, randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To maintain the blinding of the study drug (BoNT-A or placebo), all study personnel will be blinded to subjects' treatment assignment. Physicians, nurses, subjects, and any study personnel performing assessments must NOT be informed of the subject's treatment assignment except in the event of a medical emergency or as required by regulatory authorities. The injection syringes will be prepared by pharmacy personnel not involved in the study to ensure that the clinical site staff responsible for administering the study drug and conducting assessments per the protocol, and the subject, remain blinded to study treatment. Moreover, the BoNT-A and placebo solution will be limpid and indistinguishable, to maintain blindness. Both subjects, investigators and study personnel will maintain blindness to the treatments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: BoNT-A arms (Experimental): Subjects randomized in experimental group will receive intradermal injections of BoNT-A into the wrist and skin area of the hand where the pain is located.
  Interventions: Drug: BoNT-A
- Control group: Placebo arms (Placebo Comparator): Subjects randomized in control group will receive intradermal injections of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BoNT-A — A vial of 500 units of BoNT-A will be reconstituted with 2 mL of saline solution (0.9%) and 1 mL of lidocaine solution (2%) to obtain a final concentration of BoNT-A of 166.6 units/mL.
  Injections will be repeated at sites 1-1.5 cm apart (0.1 ml, 16.6 units per site), up to 20 sites (333 units).
  To reduce pain caused by the injection, lidocaine and prilocaine cream will be applied to the skin area 60 min before the procedure. Additionally, ice could be applied for a few seconds (4-8) before each injection of 16.6 units of BoNT-A.
  Injections will be repeated at week 0 and week 12.
  The active treatment and placebo solutions will be transparent and indistinguishable to maintain treatment blindness.
  Other Names: Experimental intervention
  Arms: Experimental group: BoNT-A arms
Drug: Placebo — Placebo will consist of equal volume of saline solution (0.9%). Injections will be repeated at sites 1-1.5 cm apart (0.1 ml, 16.6 units per site), up to 20 sites (333 units).
  To reduce pain caused by the injection, lidocaine and prilocaine cream will be applied to the skin area 60 min before the procedure. Additionally, ice could be applied for a few seconds (4-8) before each injection.
  Injections will be repeated at week 0 and week 12.
  The active treatment and placebo solutions will be transparent and indistinguishable to maintain treatment blindness.
  Other Names: Control intervention
  Arms: Control group: Placebo arms

SUMMARY:
The main purpose of the study is to assess the safety and efficacy of repeated administrations of BoNT-A in subjects with NP attributable to carpal tunnel syndrome (CTS) through a randomized, double-blind, placebo-controlled study. Further research has shown that BoNT-A has analgesic properties independently from its action on muscle tone, possibly by acting on neurogenic inflammation. Therefore, the study drug may be better than other treatments surgical or non-surgical currently available for the treatment of CTS.

DETAILED DESCRIPTION:
Botulinum toxin type A (BoNT-A) is widely used to treat muscle hyperactivity, based on its ability to inhibit synaptic exocytosis and, therefore, to disable neural transmission. Further research has shown that BoNT-A has analgesic properties independently from its action on muscle tone, possibly by acting on neurogenic inflammation. Animal studies indeed showed that botulinum neurotoxin can alter and alleviate NP in animals through several mechanisms, including blocking the release of pain mediators, decreasing local inflammation around nerve terminals, deactivating sodium channels, inhibiting the discharge of muscle spindles and decreasing sympathetic transmission.

Evidence on the use of BoNT-A in CTS and occipital neuralgia is still limited as it derives from small patient studies with controversial results, and is therefore considered still insufficient to determine whether or not BoNT-A could be part of the therapeutic arsenal against these NPs (level U). Overall, according to the litterature, the results of BoNT-A injections on NP are variable, as it seems to be effective in postherpetic neuralgia (evidence level A), may be effective in trigeminal neuralgia and post-traumatic neuralgia (level B) and is possibly effective in diabetic polyneuropathy (level C).

In this multicenter, randomized, double-blinding, placebo-controlled, parallel study it will enroll 164 subjects, both genders, aged ≥18 and ≤60 years old, to obtain 164 overall valuable subjects (23/24 for each center). The recruitment period (V1) will last 1 week after the baseline assessment, eligible subjects will be randomly assigned (1:1) to BoNT-A or placebo arm and will receive the first round of injections. After 12 week ±4 days (V2) subjects will undergo the second treatment round, receiving either a second BoNT-A administration or a second placebo administration. In week 24 ±4 days (V3) the same assessment scheduled for visit 1 will be repeated.

Benefit Assessment :

As described previously, BoNT-A showed some significant advantages over NPs existing treatments, such as the extended duration of its analgesic effects; BoNT-A has analgesic properties independently from its action on muscle tone, possibly by acting on neurogenic inflammation.

Therefore the study drug may be better than other treatments surgical or non-surgical currently available for the treatment of Carpal Tunnel Syndrome.

Risk Assessment :

Since it has been shown that BoNT-A has a clinically acceptable safety profile, there are no specific risks to this study.

However, considering that the drug has never been tested on patients with carpal tunnel syndrome, the objective of the study also includes the evaluation of its safety in the context of this disease.

Primary Objective

- The main objective of the study is to assess the efficacy and safety of two successive intradermal administrations of several injections of BoNT-A versus placebo, administered 12 weeks apart, in subjects with CTS and NP Secondary Objectives

The secondary objectives of this study include:

* Assessment of the therapeutic gain of BoNT-A in terms of relief of spontaneous pain.
* Assessment of BoNT-A effects in reducing neuropathic symptoms.
* Assessment of BoNT-A impact on patient's quality of life.
* Assessment of BoNT-A safety and tolerability

Statistical Hypotheses A sample size of 82 participants per group (164 participants overall) would be needed for 90% power to detect a mean difference in pain intensity between groups of 0.7 units (SD=1.3) in a two-sample two tailed t test with a type I error of 0.05, including a 10% of dropout rate. Changes in primary and secondary outcome measures (quantified measures of deficits and pains, pain scores, symptoms, quality of life) will be expressed as differences between baseline and the values obtained at each time point and will be analyzed using a generalized linear mixed-model repeated measures. For all the pre specified endpoints, the analysis will be performed in the intent-to treat population with both the last observation carried forward approach (primary analysis) and observed data (additional analysis- sensitivity). Safety data will be tabulated and where appropriate, analyzed using descriptive statistics. All tests will be two sided and a p-value of less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged ≥18 and ≤60 years old.
2. Probable or definitive NP according to the International Association for the Study of Pain criteria.
3. Daily pain attributable to CTS for at least 6 months. This must be attributable to idiopathic carpal tunnel syndrome and with nerve conduction velocity findings consistent with this condition
4. Moderate-severe pain according to the 11-point Numerical. Rating Scale (NRS; 4-8)
5. We allow the concomitant use of analgesic treatments if they have been used at a stable doses for 4 weeks before the enrolment and for the whole study.
6. Signed informed consent prior to participation in the study

Exclusion Criteria:

1. Pain level ≥9 on 11-point NRS.
2. CTS with atrophy of median-innervated muscles and EMG study suggesting a severe nerve injury.
3. Subject with contraindications or hypersensitivity to BoNT-A.
4. Subject with disorders of the neuromuscular junction, progressive neuropathy disorders, coagulation disorders or major psychiatric disorders.
5. Subject with diabetes, rheumatoid arthritis, connective tissue diseases, vasculitis, untreated hypothyroidism, acromegaly.
6. Subject using drugs acting on neuromuscular junctions, topical drugs (e.g., capsaicin or lidocaine), or anesthetic blocks.
7. Subject has used BoNT-A.
8. Subject is pregnant or breastfeeding women.
9. Subject enrolled in another interventional trial for the treatment of of the same disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of two successive administrations of several injections of BoNT-A, compared with placebo by NRS | 25 weeks
  The primary outcome is mesured as:
  -Change in mean weekly self-reported average daily pain intensity (mean pain over the past 24 hours recorded every morning in patient's diary during a week) measured by the 11-point numerical rating scale (NRS, 0=no pain, 10=maximum pain imaginable) of the brief pain inventory (BPI) from baseline (one week before randomisation) to 24 weeks after the first administration.
Efficacy of two successive administrations of several injections of BoNT-A, compared with placebo by NRS | 25 weeks
  The primary outcome is mesured as:
  - Change in weekly self-reported maximum daily pain intensity (maximum pain intensity over the past 24 hours recorded every morning in patient's diary) measured by the 11-point NRS (NRS, 0=no pain, 10=maximum pain imaginable) of the BPI from baseline (1 week before randomisation) to 24 weeks after the first administration.

SECONDARY OUTCOMES:
Assessment of the therapeutic gain of BoNT-A in terms of relief of spontaneous pain | 25 weeks
  Therapeutic gain of the second administration of BoNT-A in terms of relief of spontaneous pain, measured as change in mean weekly average daily pain intensity, measured by the 11-point numerical rating scale (NRS, 0=no pain, 10=maximum pain imaginable) of the BPI , and change in maximum pain in subjects who received two administrations.
Assessment of BoNT-A effects in reducing neuropathic symptoms with Bedside Sensory Assessment. | 25 weeks
  Effects of BoNT-A on
  - sensory disturbances and hyperalgesia in response to mechanical punctate and thermal stimuli measured by sensory assessment at the bed side; The subject examined at the bed side describes the sensation after a precise and reproducible stimulus is applied. To assess either a loss (negative sensory signs) or a gain (positive sensory signs) of somatosensory function, the responses are graded as normal, decreased or increased.
  The stimulus evoked (positive) pain types are classified as hyperalgesic (experiencing increased pain from a stimulus that is normally perceived as less painful) or allodynic (experiencing pain from a stimulus that does not normally trigger a pain response), and according to the dynamic or static character of the stimulus.
Assessment of BoNT-A effects in reducing neuropathic symptoms with VAS. | 25 weeks
  Effects of BoNT-A on
  - severity of brush-induced allodynia measured by a brush on the Visual Analogue Scale, a self-reported scale consisting of a horizontal or vertical line, usually 10 centimetres long (100 mm) anchored at the extremes by two verbal descriptors referring to the pain status.
Assessment of BoNT-A effects in reducing neuropathic symptoms with the Neuropathic Pain Symptom Inventory . | 25 weeks
  Effects of BoNT-A on
  - neuropathic symptoms (ie, burning pain, deep pain, paroxysmal pain, paraesthesia or dysaesthesia, and allodynia) measured with the Neuropathic Pain Symptom Inventory (NPSI).
  This questionnaire rates the intensity of five neuropathic dimensions (symptom combinations) during the last 24 hours (burning, deep pain, paroxysmal pain, allodynia/hyperalgesia, paresthesia/dysesthesia) on an 11-point (0-10) numerical scale.
Assessment of BoNT-A impact on patient's quality of life. | 25 weeks
  Impact of BoNT-A treatment on patient's quality of life, measured through Visual Analogue Scale of the 5-level EuroQoL (EQ-5D-5L) from 0 (imaginable health state) to 100 (worst imaginable health state) at baseline and after 24 weeks.
Assessment of BoNT-A safety | 24 weeks
  BoNT-A's overall safety and tolerability will be assessed throughout the study by measuring the occurrence and grade of AEs or serious AEs (SAEs), both registered by the subject in the patient diary or assessed by the physician during the visit(s). All AEs will be identified using MedDRA terms and will be evaluated for intensity and correlation with treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Aou Mater Domini, Catanzaro, Italy

REFERENCES:
- [Result] Attal N, de Andrade DC, Adam F, Ranoux D, Teixeira MJ, Galhardoni R, Raicher I, Uceyler N, Sommer C, Bouhassira D. Safety and efficacy of repeated injections of botulinum toxin A in peripheral neuropathic pain (BOTNEP): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2016 May;15(6):555-65. doi: 10.1016/S1474-4422(16)00017-X. Epub 2016 Mar 2. PMID 26947719
- [Result] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Result] Brown EA, Schutz SG, Simpson DM. Botulinum toxin for neuropathic pain and spasticity: an overview. Pain Manag. 2014 Mar;4(2):129-51. doi: 10.2217/pmt.13.75. PMID 24641437
- [Result] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Result] Colloca L, Ludman T, Bouhassira D, Baron R, Dickenson AH, Yarnitsky D, Freeman R, Truini A, Attal N, Finnerup NB, Eccleston C, Kalso E, Bennett DL, Dworkin RH, Raja SN. Neuropathic pain. Nat Rev Dis Primers. 2017 Feb 16;3:17002. doi: 10.1038/nrdp.2017.2. PMID 28205574
- [Result] Geoghegan JM, Clark DI, Bainbridge LC, Smith C, Hubbard R. Risk factors in carpal tunnel syndrome. J Hand Surg Br. 2004 Aug;29(4):315-20. doi: 10.1016/j.jhsb.2004.02.009. PMID 15234492
- [Result] Hobson-Webb LD, Juel VC. Common Entrapment Neuropathies. Continuum (Minneap Minn). 2017 Apr;23(2, Selected Topics in Outpatient Neurology):487-511. doi: 10.1212/CON.0000000000000452. PMID 28375915
- [Result] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Result] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Result] Marti C, Hensler S, Herren DB, Niedermann K, Marks M. Measurement properties of the EuroQoL EQ-5D-5L to assess quality of life in patients undergoing carpal tunnel release. J Hand Surg Eur Vol. 2016 Nov;41(9):957-962. doi: 10.1177/1753193416659404. Epub 2016 Jul 20. PMID 27435748
- [Result] Middleton SD, Anakwe RE. Carpal tunnel syndrome. BMJ. 2014 Nov 6;349:g6437. doi: 10.1136/bmj.g6437. No abstract available. PMID 25378457
- [Result] Mittal SO, Safarpour D, Jabbari B. Botulinum Toxin Treatment of Neuropathic Pain. Semin Neurol. 2016 Feb;36(1):73-83. doi: 10.1055/s-0036-1571953. Epub 2016 Feb 11. PMID 26866499
- [Result] Olney RK. Carpal tunnel syndrome: complex issues with a "simple" condition. Neurology. 2001 Jun 12;56(11):1431-2. doi: 10.1212/wnl.56.11.1431. No abstract available. PMID 11402097
- [Result] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Result] Ranoux D, Attal N, Morain F, Bouhassira D. Botulinum toxin type A induces direct analgesic effects in chronic neuropathic pain. Ann Neurol. 2008 Sep;64(3):274-83. doi: 10.1002/ana.21427. PMID 18546285
- [Result] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Result] Attal N, Fermanian C, Fermanian J, Lanteri-Minet M, Alchaar H, Bouhassira D. Neuropathic pain: are there distinct subtypes depending on the aetiology or anatomical lesion? Pain. 2008 Aug 31;138(2):343-353. doi: 10.1016/j.pain.2008.01.006. Epub 2008 Mar 4. PMID 18289791